CLINICAL TRIAL: NCT03978234
Title: A Phase II Clinical Trial Evaluating the Safety and Effect of abobotulinumtoxinA Injection in the Gastrocnemius Muscle to Improve Equinus and Associated Plantar Fasciitis Pain
Brief Title: Evaluating the Safety and Effect of abobotulinumtoxinA in the Gastrocnemius Muscle to Improve Equinus and Plantar Fasciitis Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Foot and Ankle Foundation (Other)
Responsible Party: Principal Investigator, Maha K. Curley, Study Coordinator, University Foot and Ankle Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFAI-PF-01
Record Dates: First submitted 2019-05-23; First posted 2019-06-07 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Plantar Fasciitis; Plantar Fasciitis, Chronic; Plantar Fasciitis of Both Feet
Keywords: Heel pain; Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): Single group
  Interventions: Drug: AbobotulinumtoxinA 300 UNT

INTERVENTIONS:
Drug: AbobotulinumtoxinA 300 UNT — AbobotulinumtoxinA 300 UNT

SUMMARY:
The purpose of this research is to collect safety and efficacy data on injection of botulinumtoxinA (AbobotulinumtoxinA /Dysort) into the gastrocnemius (calf) muscle to improve equinus (lack of flexibility to bring the top of the foot towards the front of the leg) in subjects with plantar fasciitis and relieve pain associated with this condition. The use of AbobotulinumtoxinA is considered experimental in this study because it has not been approved by the United States Food and Drug Administration (FDA) for the treatment of plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old and not older than 75 years.
2. History of Plantar fasciitis for a minimum of 6 weeks
3. History and physical examination consistent with plantar fasciitis and a diagnostic ultrasound study showing thickening of the plantar fascia >5 mm (normal is 3 mm)
4. Minimum Visual Analog Scale (VAS) score of 4.
5. Failed conservative care with at least two of the following treatments: Stretching, rest, shoe modifications, insoles or orthotics, physical therapy, or cortisone injection.
6. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
7. Subject understands and is willing to participate in the clinical study and can comply with visit and post -injection questionnaire schedules.

Exclusion Criteria:

1. Patients with history of diabetes, back issues, nerve issues or previous surgery of the foot or calf.
2. Patients with no pain in the heel region.
3. Subject is pregnant or breast- feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
injection | 8 weeks
  Reduction of pain (VAS scale) associated with plantar fasciitis at 8 weeks post injection

SECONDARY OUTCOMES:
Adverse Events | 26 weeks
  Number of product related AEs per patient that are definitely, probably, or possibly related to the product post-injection
PROMIS Pain intensity instrument | 26 weeks
  Changes in PROMIS Pain Intensity Instrument,
PROMIS Pain interference instrument | 26 weeks
  Changes in PROMIS Pain Interference Instrument
PROMIS Physical function Instrument | 26 weeks
  Changes in PROMIS Physical function instrument
AOFAS Ankle-Hindfoot Score | 26 weeks
  Changes in the American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Score
FAAM Foot and Ankle Ability Measure | 26 weeks
  Changes in the Foot and Ankle Ability Measure
Gastrocnemius measurement | 26 weeks
  Changes in gastrocnemius muscle size using ultrasonography
Gastrocnemius measurement and mobility | 26 weeks
  Changes in gastrocnemius range of motion/dorsiflexion using goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Babak Baravarian, DPM, Principal Investigator — University Foot & Ankle Foundation
Locations (1):
- University Foot & Ankle Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://footankleinstitute.com